CLINICAL TRIAL: NCT01058902
Title: The Effect Of Aspirin On Survival Following Potentially Curative Resection Of Non Small Cell Carcinoma Of The Lung The Big A Trial
Brief Title: The Effect Of Aspirin On Survival in Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: failed to achive funding
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Mike Poullis, Consultant Cardiothoracic Surgeon, Liverpool Heart and Chest Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-018360-16
Record Dates: First submitted 2010-01-26; First posted 2010-01-29 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Non Small Cell Lung Cancer; Survival; Aspirin
Keywords: Non small cell lung cancer; survival; aspirin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Aspirin; N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Negative control (Placebo Comparator): Not on aspirin pre operatively, but refuse to enter trial or have a contraindication to aspirin
  Interventions: Other: no aspirin
- Aspirin treatment (Experimental): group randomised to aspirin
  Interventions: Drug: Aspirin 75 mg
- No aspirin treatment (Experimental): Randomised to no aspirin
  Interventions: Other: no aspirin
- Positive control (Active Comparator): Already on aspirin. just observational limb
  Interventions: Drug: Aspirin 75 mg

INTERVENTIONS:
Drug: Aspirin 75 mg — Aspirin 75 mg
  Other Names: PL 00142/0377 Activis
  Arms: Aspirin treatment; Positive control
Other: no aspirin — nothing
  Other Names: Observation of patients on their pre op medications
  Arms: Negative control; No aspirin treatment

SUMMARY:
Lung cancer is the most common cancer in the western world. Only 10 to 15 % of patients diagnosed with lung cancer are suitable for potentially curative surgical treatment. Despite surgery, recurrence of lung cancer still occurs. Aspirin potentially may help increase survival by altering the biochemistry of any potential remaining lung cancer cells. Most lung cancer occurs in smokers. Smokers are at increased risk of heart attacks and strokes. Aspirin has beneficial effects on the heart and brain, potentially reducing the incidence of heart attacks and strokes.

DETAILED DESCRIPTION:
Study design Randomised study of aspirin 75mg to reduce the mortality in patients after resection of non-small cell lung cancer. Patients already on aspirin, unsuitable for study or not wishing to partake in this study will be asked for permission to be followed up via their GP and the National Strategic Tracking service.

Methodology Initially all consultant thoracic and cardiothoracic surgeons in the UK will be consulted to obtain permission for their patients to be included in this study. If they agree the individual units' lung cancer nurses will actually be involved in recruiting post operative patients into the study. We will use the lung cancer nurses to enter via a secure electronic system patients pre operative characteristics and post operative staging and histology. Mortality will followed via the strategic tracing service.

Study subjects/patients All patients undergoing potentially curative resection of non small cell carcinoma of the lung. Patients will be recruited post operatively so that post operative deaths are eliminated, and histology is known prior to randomisation.

Contamination of control limb

Patients in the aspirin limb will be asked at their 1 year, 3 years and 5 years out patient appointment if they are still staking the aspirin. Patients in the control limb will be asked at their 1 year, 3 years and 5 years out patient appointment if they have been started on aspirin by anyone.

If these appointments are missed the patients GP will be contacted for this information, as long as the patient has agreed for us to contact their GP.

Data collection This will be prospective via a secure web server, hosted on an NHS computer located in a secure NHS IT locked room.

Study procedures No invasive procedure, samples or tissues will be performed or obtained in any patients.

Study intervention Aspirin 75 mg/day or no tablet taken for a period of 5 years after randomisation.

Reducing adverse events

All patients will be assessed by the researcher to eliminated patients with as history of gastric or duodenal ulcers, or known allergy to aspirin or other NSAIDs.

Monitoring of Adverse events All patients will be given a business card with a contact number, an email address and a web address so that they can report all adverse events while participating in this trial. In addition all general practitioners with patients in the trial will be notified.

Specific adverse events we will be following include:

Stopping trial medication secondary to side effects, GI bleeds, stomach ulcers, anaemia that require hospital admission and Blood transfusion(s)

Data Monitoring Committee The data management committee will analyse survival data in the control and intervention limb every 6 months up to 5 years with regard to mortality and gastrointestinal side effects that required hospital admission.

If the mortality in the aspirin treatment group exceeds more than 3 Standard deviations above the control mortality rate the trial will be stopped immediately and the aspirin users all contacted immediately and informed to stop the aspirin immediately.

The gastrointestinal side effects of aspirin have been widely studied and as aspirin is an over the counter product being used in its lowest dose formulation we do not aim to use gastrointestinal side effects as a marker for stopping the trial.

GP contacts All GPs will be informed of their patients inclusion in this trial.

Statistical analysis. This will be performed by Dr Mark Jackson or a delegated member of his team, at Liverpool Heart and Chest Hospital.

Sample size Based on a retrospective trail conducted in Liverpool Heart and Chest hospital. Accepting the suggested hazard ratio of 0.84 and a difference in 5-year survival of approximately 6%, various power calculations were performed to derive an estimate of the sample size required for such a trial. Depending on the aspirin:non-aspirin ratio and based on standard assumptions, a combined total of between 2000 and 3000 patients would need to be recruited to detect a significant difference in survival. Hence we aim to recruit 2,500 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 to 85, undergoing potentially curative resection of non small cell carcinoma of the lung, who have none of the following exclusion criteria.

Exclusion Criteria:

* Already on aspirin Small cell carcinoma N2 disease Confirmed metastatic disease Incomplete resections Previous cancer in last 3 years History of gastric or duodenal ulcers Known allergy to aspirin or other NSAIDs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Survival - alive or dead (A standard cancer trial outcome). This will be assessed via the UK national strategic tracking service | 5 years

SECONDARY OUTCOMES:
Side effects eg gastrointestinal | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mike Mr Poullis, FRCS(CTh), Principal Investigator — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, Merseyside, United Kingdom